CLINICAL TRIAL: NCT02253420
Title: An Open-label Non-randomized, Phase 1 Study to Evaluate the Effect of (a) Itraconazole or Rifampin on the Pharmacokinetics of a Single Intravenous Dose of Copanlisib and (b) Copanlisib on Cardiovascular Safety in Subjects With Advanced Solid Tumors and Non-Hodgkin's Lymphoma
Brief Title: COPANLISIB (BAY80-6946) Drug-drug Interaction and Cardiovascular Safety Study in Advanced Solid Tumor and Non-Hodgkin's Lymphoma Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 16270
Record Dates: First submitted 2014-09-29; First posted 2014-10-01 (Estimated); Last update posted 2020-12-14 (Actual); Status verified 2020-12

CONDITIONS: Medical Oncology
Keywords: Phase 1; Advanced solid tumor; non-Hodgkin's lymphoma; PI3 Kinase inhibitor; Drug-drug Interaction
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — copanlisib; Itraconazole; Rifampin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Copanlisib with and without concomitant Itraconazole (Arm A) (Experimental): To evaluate the effect of Itraconazole on the pharmacokinetics of Copanlisib (BAY80-6946) and safety in patients with advanced solid tumor. Cycle 1 of the study will be conducted in 2 parts: Part 1 and part 2:
  * Part 1 of Cycle 1: 6 patients will be enrolled and will receive 12 mg of copanlisib on Day 1 and Day 15. Itraconazole 200 mg will be administered twice a day on Day 12 and then once daily from Days 13 to 21.
  * Part 2 of Cycle 1: 20 patients will be enrolled and receive copanlisib doses of either 12 mg, 30 mg or 60 mg on Days 1 and 15 with the same dose administered on both days. Copanlisib dose for Part 2 will be based on safety and copanlisib pharmacokinetics in Part 1. Itraconazole 200 mg will be administered twice a day on Day 12 and then once daily from Days 13 to 21.
  * Cycle 2 and subsequent cycles: All patients will receive copanlisib doses of 60 mg on Days 1, 8 and 15.
  Interventions: Drug: Copanlisib (BAY80-6946); Drug: Itraconazole
- Copanlisib with and without concomitant Rifampin (Arm B) (Experimental): To evaluate the effect of Rifampin on the pharmacokinetics of Copanlisib (BAY 80-6946) and safety in patients with advanced solid tumor or non-Hodgkin's lymphoma in Cycle 1. Approximately 30 subjects will receive 60mg of copanlisib on Cycle 1 Day 1 and Cycle 1 Day 15. Rifampin will be administered once a day from Cycle 1 Day 10 to Day 21. Holter monitoring will be performed on Cycle 1 Day -1 and Cycle 1 Day 1 to evaluate the effect of copanlisib on the QT/QTc assessment.
  Cycle 2 and subsequent cycles, all patients will receive copanlisib dose of 60 mg on Days 1, 8 and 15. Holter monitoring will be performed on Cycle 3 Day 1 and Cycle 6 Day 1.
  Interventions: Drug: Rifampin; Drug: Copanlisib (BAY80-6946)

INTERVENTIONS:
Drug: Copanlisib (BAY80-6946) — Part 1 of Cycle 1 Cycle 1 Day 1: Single i.v. dose 12mg Cycle 1 Day 15: Single i.v. dose 12 mg Part 2 of Cycle 1 Cycle 1 Day 1: Single i.v. dose 60mg (based on Part 1 data) Cycle 1 Day 15: Single i.v. dose 60mg (based on Part 1 data)
  Part 1 & Part 2
  Cycle 2 and subsequent cycles:
  Day 1: Single i.v. dose of 60mg Day 8: Single i.v. dose of 60mg Day15: Single i.v. dose of 60mg
  Arms: Copanlisib with and without concomitant Itraconazole (Arm A)
Drug: Itraconazole — Cycle 1 Day 12: 2 x 200 mg itraconazole oral (two doses, 12 hours apart) Cycle 1 Days 13-21: 200 mg itraconazole oral, once daily in the morning
  Arms: Copanlisib with and without concomitant Itraconazole (Arm A)
Drug: Rifampin — Cycle 1 Days 10 - 21: 600mg Rifampin oral, once daily in the morning
  Arms: Copanlisib with and without concomitant Rifampin (Arm B)
Drug: Copanlisib (BAY80-6946) — Cycle 1 Day 1: Single i.v. dose 60mg Cycle 1 Day 15: Single i.v. dose 60mg
  Cycle 2 and subsequent cycles:
  Day 1: Single i.v. dose of 60mg Day 8: Single i.v. dose of 60mg Day15: Single i.v. dose of 60mg
  Arms: Copanlisib with and without concomitant Rifampin (Arm B)

SUMMARY:
To evaluate the effect of itraconazole or rifampin on the absorption, distribution, metabolism and elimination of COPANLISIB (BAY80-6946).

To evaluate the effect of copanlisib on QT/QTc intervals and left ventricular ejection fraction as parameters of cardiovascular safety.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients ≥ 18 years of age with histological or cytological confirmed advanced solid tumors or non-Hodgkin's lymphoma that have progressed on, or failed to respond to, therapies known to provide clinical benefit may be enrolled after signing informed consent.
* Normal left ventricular ejection fraction; adequate liver, renal and bone-marrow functions as assessed by laboratory values.
* Adequate performance status and life expectancy of at least 3 months.

Exclusion Criteria:

* Solid-tumor patients with central nervous system (CNS) metastases if treatment completed < 3 months before enrollment or lesions unstable or progressing on MRI scans performed within 1 month of enrollment or unstable symptoms of the CNS metastases.
* Evidence of ventricular dysfunction such as congestive heart failure (CHF) or a history of CHF greater than NYHA Class II
* Active coronary artery disease or myocardial infarction within the 6 months before study entry; any new-onset angina within the 3 months before study entry or unstable angina; cardiac arrhythmia requiring anti-arrhythmic therapy.
* Prior diagnosis of Type 1 or 2 diabetes mellitus, hyperglycemia (defined as fasting blood or plasma glucose above 125 mg/dL under 2 separate days, corresponding to 6.94 mmol/L) or HbA1c ≥ 7%.
* Use of systemic including inhaled corticosteroids within the 2 days before the start of study treatment (however, topical steroids are permitted).
* Known presence of human immunodeficiency virus (HIV) infection or active hepatitis (B or C).
* Uncontrolled hypertension (systolic blood pressure [BP] >150 mmHg or diastolic blood pressure > 90 mmHg despite optimal medical management).
* Anticancer chemotherapy, hormone therapy or immunotherapy within the 4 weeks before the first study treatment or scheduled for administration (of the above) during the study
* History of, or concurrent, interstitial lung disease (ILD) or severely impaired pulmonary function.
* Medications with drug-drug interaction potential for itraconazole which is to be excluded before the study and during Cycle 1 such as CYP3A4 substrates with a narrow therapeutic window or which have the potential to prolong QTc
* Concomitant medication contraindicated for use with rifampin (including, but not limited to): cisapride, oral midazolam, nisoldipine, pimozide, quinidine, dofetilide, triazolam, levacetylmethadol (levomethadyl), 3-hydroxy-3-methyl-glutaryl coenzyme A (HMG-CoA)-reductase inhibitors metabolised by CYP3A4, such as lovastatin and simvastatin, ergot alkaloids metabolised by CYP3A4, such as dihydroergotamine, ergometrine (ergonovine), ergotamine and methylergometrine (methylergonovine), atazanavir, darunavir, fosamprenavir, ritonavir-boosted saquinavir, saquinavir, or tipranavir

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2014-10-08 (Actual); Primary Completion 2018-03-12 (Actual); Study Completion 2019-08-13 (Actual)

PRIMARY OUTCOMES:
AUC (0-168) | Within cycle 1, at pre-dose and at 10 min, 1, 1.33 (arm B)1.5 (arm A), 2, 2.5, 3, 5, 8, 24, 48, 72, 96, 120, and 168 hours after start of drug infusion on Days 1 and 15.
  AUC (0-168): Area under the curve from dosing to 168 h after dosing
AUC | Within cycle 1, at pre-dose and at 10 min, 1, 1.33 (arm B)1.5 (arm A), 2, 2.5, 3, 5, 8, 24, 48, 72, 96, 120, and 168 hours after start of drug infusion on Days 1 and 15.
  AUC: Area under the curve
Cmax | Within cycle 1, at pre-dose and at 10 min, 1, 1.33 (arm B)1.5 (arm A), 2, 2.5, 3, 5, 8, 24, 48, 72, 96, 120, and 168 hours after start of drug infusion on Days 1 and 15.
  Cmax: Maximum concentration attained after dosing
QTcF | Holter Monitoring performed on Cycle 1 Day -1 (baseline) and Cycle 1 Day 1 (each cycle is 28 days)
  QTcF: Time-matched largest change of QT interval (Frederica's correction)

SECONDARY OUTCOMES:
AUC(0-tlast) | Within cycle 1, at pre-dose and at 10 min, 1, 1.33 (arm B)1.5 (arm A), 2, 2.5, 3, 5, 8, 24, 48, 72, 96, 120, and 168 hours after start of drug infusion on Days 1 and 15.
  AUC(0-tlast): Area under the curve from dosing to last measurable concentration
tmax | Within cycle 1, at pre-dose and at 10 min, 1, 1.33 (arm B)1.5 (arm A), 2, 2.5, 3, 5, 8, 24, 48, 72, 96, 120, and 168 hours after start of drug infusion on Days 1 and 15.
  tmax: Time from dosing to attainment of Cmax
tlast | Within cycle 1, at pre-dose and at 10 min, 1, 1.33 (arm B)1.5 (arm A), 2, 2.5, 3, 5, 8, 24, 48, 72, 96, 120, and 168 hours after start of drug infusion on Days 1 and 15.
  tlast: Time from dosing to last measurable concentration
t1/2 | Within cycle 1, at pre-dose and at 10 min, 1, 1.33 (arm B)1.5 (arm A), 2, 2.5, 3, 5, 8, 24, 48, 72, 96, 120, and 168 hours after start of drug infusion on Days 1 and 15.
  t1/2: Terminal half-life
Urine [AE,ur(0-24)] | From 0-8 hours and >8 up to 24 hours after the start of copanlisib infusion on Days 1 and 15 of Cycle 1
  Amount of drug excreted via urine during the collection interval 0 - 24 hours post administration
Number of participants with adverse events as a measure of safety and tolerability | At approximately 29 months
  Safety analysis will be conducted continuously until safety follow-up
PR intervals | Holter Monitoring performed on Cycle 1 Day -1 (baseline) and Cycle 1 Day 1 (each cycle is 28 days)
QRS intervals | Holter Monitoring performed on Cycle 1 Day -1 (baseline) and Cycle 1 Day 1 (each cycle is 28 days)
ECG waveform morphology | Holter Monitoring performed on Cycle 1 Day -1 (baseline) and Cycle 1 Day 1 (each cycle is 28 days)
Left ventricular ejection fraction (LVEF) | At baseline, in the last week of Cycle 1, and in the last 2 weeks of Cycle 2, Cycle 3, Cycle 6 and every third cycle (Cycle 9, Cycle 12, etc.) and end of treatment
  MUGA scans
QTcB | Holter Monitoring performed on Cycle 1 Day -1 (baseline) and Cycle 1 Day 1 (each cycle is 28 days)
  QTcB: Bazett's corrected QT interval

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (5):
- Dallas, Texas, United States
- Canada (4):
  - Edmonton, Alberta
  - Vancouver, British Columbia
  - Hamilton, Ontario
  - Toronto, Ontario

IPD SHARING:
Plan to Share IPD: Undecided
Availability of this study's data will be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access.
  As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.clinicalstudydatarequest.com to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the Study sponsors section of the portal.